CLINICAL TRIAL: NCT04118543
Title: Oxfordshire Sedentariness, Obesity & Cardiometabolic Risk in Adolescents - a Trial of Exercise in Schools
Acronym: OxSOCRATES
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Oxford (Other)
Collaborators: Oxford Brookes University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: R54302/RE001
Record Dates: First submitted 2019-09-04; First posted 2019-10-08 (Actual); Last update posted 2021-08-12 (Actual); Status verified 2021-08

CONDITIONS: Overweight/Obesity, Adolescent
Keywords: Obesity; Cardiometabolic; Adolescence; Exercise
MeSH Terms: conditions — Overweight; Obesity; Motor Activity

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): The intervention group will take part in three 1-hour targeted moderate-to-vigorous physical activity (MVPA) gym-based group exercise sessions per week for eight weeks with individualised prescriptions.
  Interventions: Other: Intervention Group
- Sham-Exercise Group (Sham Comparator): The shame-exercise group will complete three sham exercise group sessions per week for eight weeks (including stretching, coordination and balance activities and very low-level cardiovascular activities that mimic the types of exercise done in the intervention group).
  Interventions: Other: Sham-Exercise Group

INTERVENTIONS:
Other: Intervention Group — Each participant assigned to this intervention arm will start with a progressive cardiovascular warm-up for 10mins. The main exercise session will consist of resistance and cardiovascular based exercises targeting the whole body, which will last for 35-40mins. A cool-down period will follow lasting 5-10mins.
  Other Names: Exercise Intervention Group
  Arms: Intervention Group
Other: Sham-Exercise Group — Each participant assigned to this intervention arm will start with a warm-up for 10mins, which will be controlled in order to reduce any cardiovascular training effects. The sham-exercise sessions will consist of stretching, coordination and balance activities and very low-level cardiovascular activities that mimic the types of exercise done in the intervention group. This will last for 35-40mins, followed by a 5-10min cool-down.
  Arms: Sham-Exercise Group

SUMMARY:
Obesity is a major cardiovascular disease (CVD) risk factor that is rising fastest in children. Prevention of its damaging effects should begin earlier before they become irreversible. Pilot data identified novel markers of cardiometabolic dysfunction that may be better than body mass index at stratifying risk and as targets for CVD prevention in the young. Advanced imaging, blood tests and a meal-challenge will be used to comprehensively characterise how early metabolic dysfunction (liver and muscle fat, insulin resistance) affects cardiovascular health (arterial stiffness, myocardial energetics, gut vasoreactivity, diastolic function, blood pressure trajectory, left ventricular hypertrophy) in 210 adolescents (110 obese, 50 sedentary normal-weight, 50 high-activity). Reversibility of this phenotype will be tested in the obese by randomised controlled trial, comparing 8-week supervised exercise to a low-activity sham intervention. This study will provide the platform for developing practical, effective CVD prevention in children that is not simply focused on weight-loss.

DETAILED DESCRIPTION:
Objectives and Outcome measures

This proposal aims to (1) improve identification of early cardiometabolic dysfunction in children and (2) investigate the reversibility of this dysfunction through exercise. The study will provide the platform for developing practical, effective primordial CVD prevention strategies and the identification of novel early therapeutic targets.

Study Design

This study combines elements of both observational and interventional study designs. A prospective, cross-sectional study of adolescents with 1-year follow-up is combined with a randomised placebo (sham-exercise)-controlled trial (RCT) of eight-weeks of supervised, individualised exercise in an obese sub-population. The RCT is of an established, standardised exercise programme that is low-risk. Group allocation will be known only to the exercise physiologist and staff carrying out the exercise intervention.

Fitness tests will be carried out in schools and in our exercise laboratory, which will provide opportunities to support questionnaire completion, fit accelerometers, fit and return ambulatory blood pressure monitors and address participant questions or concerns. In addition, participants will visit The Oxford Centre for Clinical Magnetic Resonance Research (OCMR) for the initial assessment and for the follow-up assessment for those participants in the obese group.

Participants

210 participants will be recruited, 110 of these will be obese, 50 will be normal weight and their activity will be matched to the obese group and therefore, relatively sedentary. 50 normal weight controls will be selected on the basis of high levels of physical activity. The 110 obese participants will be randomised (1:1) to exercise intervention or a low-intensity sham exercise placebo intervention. These numbers are justified by a priori power calculations and take into account potential withdrawals at an attrition rate of 10% that is compatible with recent studies in the same or similar populations (e.g. Fit to Study). Compliance with the interventions will be increased by carrying out the interventions through an online remote methodology which can also be implemented in a school setting, predominantly during mandatory physical education (PE) lessons. Trained, experienced staff will supervise the exercise sessions, ensuring participant engagement with the activities by measuring heart rate and physical activity levels.

Recruitment

Pre-screening will be done through schools who will write to families informing them that their children will be taking part in an enhanced P.E. lesson at school that includes a fitness and health screening session. As part of this, the children will be asked to wear an activity watch (accelerometer) for a week. The session will explore many aspects of their agility and fitness and assess their muscle strength, power, motor skills, speed, endurance and flexibility, adjusted for their physical size (height and weight). The lesson will be educational, giving personalised feedback to the children on their strengths and how to improve on areas where they are less strong. The school will retain a file linking the children's names to random identifiers but the researchers will not have access to, or retain, any identifiable information. Parents will be sent a letter giving them the opportunity to withdraw their children from this health screening session and explaining that researchers may ask the school to contact them again on their behalf if their children are eligible for study participation on the basis of their fitness assessment. Children who are withdrawn by their parents will participate in their usual P.E. lesson.

Recruitment will be done by letters to parents, delivered via the schools. Recruitment from an established population already in contact with the investigators research group should increase participation rates. It is difficult to precisely estimate the proportion of participants who fulfil the inclusion/exclusion criteria but it is assumed an obesity rate (BMI z-score (WHO) > 2) of approximately 20%.

In addition to the school screening recruitment, participants may also volunteer to take part in the study through our online advertisement and social media campaign. Children who express an interest will be invited to contact the study team so that an initial health assessment can be completed and an information pack can be provided. This pack will contain participant information sheets and consent forms, and will collect information needed for BMI z-score calculation. Then potentially eligible participants will be invited to complete physical activity questionnaires to determine eligibility and group allocation. This is to avoid any unnecessary testing on ineligible participants at university sites and provides a suitable remote method to differentiate between active and inactive participants.

Screening

Pre-stratification of the potential population for recruitment will be carried out, based on BMI and activity levels. Obese and normal weight groups will be approached for recruitment sequentially, according to their rank position within their respective BMI-based criteria in order to maximise the difference between groups (e.g. the most obese will be approached first for the obese group). The normal weight group will be further stratified according to activity levels such that half of this group matches the obesity group for activity whilst the other half are highly-active individuals. Again, individuals within this subgroup will be approached according to their rank position in the distribution of activity such that the most active are preferred in order to maximise the difference between groups.

Informed Consent

Participant's parents/guardians will be asked to sign and date the latest approved version of the Informed Consent before any study-specific procedures are performed. The latest approved Participant Information sheet will be provided to them and verbal explanations will also be provided ensuring that all of the following information has been presented and understood: the exact nature of the study; what it will involve for the participant; the implications and constraints of the protocol; and all known risks or benefits involved in taking part.

Participants will be told that they are free to withdraw from the study at any time and for any reason without being required to give a reason for their withdrawal. The participant will be allowed as much time as they wish to consider the information, and the opportunity to question the Investigator, their General Practitioner (GP) or other independent parties to decide whether they will participate in the study. Once these conditions are satisfied, written Informed Consent will be obtained by means of participant dated signature and dated signature of the person who presented and obtained the Informed Consent. The person taking consent will be a qualified member of the study team with a complete understanding of the study and with the authorisation of the Principal Investigator. A copy of the signed Informed Consent will be given to the participant and the original signed form will be retained at the study site.

Randomisation

Random allocation of members of the obese group to a sham fitness intervention or to a standardised exercise intervention will be carried out using an online randomisation process. The analysis will be carried out on an "intention-to-treat" basis when participants do not complete all elements of the data collection process and single-blinding will be maintained such that members of the team carrying out procedures at OCMR e.g. MRI and those involved in the data analysis are blinded to the allocation of intervention and sham groups. All data acquired at OCMR will be identified by a unique study number only. Inadvertent un-blinding will result in the exclusion of that individual's data from the analysis.

Incidental findings

Cardiovascular findings will be dealt with by the PI or another MRI-trained Consultant Paediatric Cardiologist. Findings in other imaging will be reviewed by the study Paediatric Radiologist. OCMR standard operation procedures (SOPs) for dealing with cardiac and non-cardiac incidental findings, respectively will be followed. Participants will not be informed of incidental findings on the day and will only be contacted after they have been formally reviewed and if a concern remains that further investigation is required.

Discontinuation or withdrawal of participants from the study

Each participant will have the right to withdraw from the study at any time. In addition, participation in the study may be discontinued at any time if the Investigator considers it necessary for any reason, including but not limited to: Pregnancy, ineligibility (either arising during the study or retrospectively, having been overlooked at screening), a significant protocol deviation, significant non-compliance with the exercise regimen or other study requirements, withdrawal of consent, and loss to follow-up. Data gathered to that point will be included in the analysis under an intention-to-treat principle. Where possible, further recruitment will be carried out to compensate for data loss resulting from early discontinuation of participation. The reason for all withdrawals will be recorded in the Case Report Form.

Confounding Factors

The exercise intervention RCT will be carried out over 8 weeks. The MRI scan operator will be blinded to RCT group allocations and all analyses will be carried out on anonymised data. Confounding factors in the observational part of the study will be addressed by matching of groups for age, sex, height, pubertal status and by matching the normal-weight sedentary group on activity level with the obese group. Questionnaires on cardiometabolic risk factors such as diet and sedentary behaviour will be used to quantify potential confounders. At least 24 hours prior to study visits, participants will be asked to avoid strenuous exercise, not smoke or drink alcohol, and eat a standardised evening meal before fasting in the morning.

Analysis

Analyses in the RCT will be carried out on an "intention-to-treat" basis. Secondary exploratory analysis will be to explore mechanisms

ELIGIBILITY:
Inclusion Criteria:

* Participants willing and able to register their informed assent and whose parent(s)/guardian(s), give informed consent for participation of their child in the study
* Age and sex-appropriate BMI scores using the World Health Organisation standards for obesity and normal weight
* Objectively measured physical activity

Exclusion Criteria:

* Contraindications for exercise intervention as determined by the Physical Activity Readiness Questionnaire
* Safety issues due to behavioural/intellectual limitations
* Medical Conditions such as neurological disorders or uncontrolled epilepsy
* Allergies to dairy
* Type 1 diabetes
* Pregnancy
* Contraindications for Magnetic Resonance scans

Ages: 11 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 210 (Estimated)
Dates: Start 2019-10-01 (Actual); Primary Completion 2023-07 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Cardiometabolic phenotype score | Changes from baseline - 8 weeks
  An additive cardiometabolic phenotype score will be defined as the sum of the z-scores of known elements of cardiometabolic risk with each element scored such that a positive value indicates greater risk.
  The following elements will be scored positively in the risk model: low cardiac phosphocreatine and adenosine triphosphate (PCr/ATP) ratio z-score by phosphate Magnetic Resonance Spectroscopy (MRS), high aortic pulse wave velocity z-score (arterial stiffness) by Magnetic Resonance (MR), high Homeostatic Model Assessment for Insulin Resistance (HOMA-IR) z-score (insulin resistance), high visceral fat mass z-score by T2*-IDEAL MR, high left ventricular mass z-score by MR, low peak left ventricular diastolic filling rate z-score by MR, and high 24 hour ambulatory blood pressure z-score.
Superior mesenteric artery blood flow after a meal challenge | Changes from baseline - 8 weeks
  Assessing the change of blood flow (l/min) in the superior mesenteric artery in response to a meal challenge, measured by phase-contrast MR.
Muscle acetylcarnitine | Changes from baseline - 8 weeks
  Increased acetylcarnitine is a marker of skeletal muscle metabolism, measured by MRS.
Triglyceride | Changes from baseline - 8 weeks
  Blood plasma (mmol/l) post prandial triglyceride response.

SECONDARY OUTCOMES:
Echocardiography - Diastolic Function | Changes from baseline - 8 weeks
  Early mitral inflow velocity and mitral annular early diastolic velocity ratio (E/E' ratio) will be derived from mitral valve inflow Doppler and Tissue Doppler Imaging of the left ventricular myocardium.
High Density Lipoprotein (HDL) | Changes from baseline - 8 weeks
  Blood samples taken at rest, measuring cholesterol (mmol/L).
Low Density Lipoprotein (LDL) | Changes from baseline - 8 weeks
  Blood samples taken at rest, measuring cholesterol (mmol/L).
Alanine aminotransferase (ALT) | Changes from baseline - 8 weeks
  Blood samples taken at rest measuring liver dysfunction (mmol/L).
Aspartate Aminotransferase (AST) | Changes from baseline - 8 weeks
  Blood samples taken at rest measuring liver dysfunction (mmol/L).
Alkaline Phosphatase (ALP) | Changes from baseline - 8 weeks
  Blood samples taken at rest measuring liver dysfunction (mmol/L).
Total Bilirubin (T.Bil) | Changes from baseline - 8 weeks
  Blood samples taken at rest measuring liver dysfunction (mmol/L).
Haemoglobin A1c (HbA1c) | Changes from baseline - 8 weeks
  Blood samples taken at rest (mmol/L).
Glucose | Changes from baseline - 8 weeks
  Serial measures after meal (mmol/L).
Insulin | Changes from baseline - 8 weeks
  Serial measures after meal (mmol/L).
Full Blood Count (FBC) | Changes from baseline - 8 weeks
  Blood samples taken at rest.
High Sensitivity C-reactive protein (CRP) | Changes from baseline - 8 weeks
  Blood samples taken at rest (mmol/L).
Food Preference Questionnaire | Changes from baseline - 4 weeks and 8 weeks
  United Kingdom (UK) Biobank Food preference Questionnaire.
Health Behaviour Questionnaire | Changes from baseline - 4 weeks and 8 weeks
  The Health Behaviour in School-Aged Children (HSBC).
Weight Related Eating Questionnaire | Changes from baseline - 4 weeks and 8 weeks
  Weight-Related Eating Questionnaire (WREQ).
Self-Regulation of Eating Behaviour Questionnaire | Changes from baseline - 4 weeks and 8 weeks
  Self-Regulation of Eating Behaviour Questionnaire (SREBQ).
Physical Activity Levels | Changes from baseline - 8 weeks
  Wrist-worn triaxial accelerometers will sample physical activity levels over seven days.
Skeletal muscle lipid | Changes from baseline - 8 weeks
  skeletal muscle lipid measured MRS.
Cardiac PCr/ATP ratio | Changes from baseline - 8 weeks
  Cardiac PCr/ATP is a measure of myocardial energetics, measure by MRS.
Cardiac lipids | Changes from baseline - 8 weeks
  Cardiac lipids is a measure of myocardial lipid spill over, measure by MRS.
Aortic pulse wave velocity | Changes from baseline - 8 weeks
  An index of arterial stiffness, measured by MR.
Homeostatic Model Assessment for Insulin Resistance (HOMA-IR) | Changes from baseline - 8 weeks
  Measures insulin resistance.
Visceral fat mass | Changes from baseline - 8 weeks
  Associated with adverse cardiometabolic changes in adolescents, measured by T2*-IDEAL MR.
Left ventricular mass | Changes from baseline - 8 weeks
  A measure of early cardiometabolic dysfunction, measured MR.
Peak left ventricular diastolic filling rate | Changes from baseline - 8 weeks
  Indicator of early cardiovascular damage, measure by MR.
Blood pressure | Changes from baseline - 8 weeks
  24 hour ambulatory systolic and diastolic blood pressure, measured by SunTech Oscar 2 monitor.
Skeletal muscle glycogen | Changes from baseline - 8 weeks
  Increased glycogen is a marker of skeletal muscle metabolism, measured my MRS.
Participant experience | At 8 weeks post baseline and 1 year follow
  Optional exit interview of study experience.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Jones, BM, BSc, FRCP, PhD, Principal Investigator — University of Oxford; Helen Dawes, PhD, Study Director — Oxford Brookes University
Locations (1):
- Oxford Centre for Clinical Magnetic Resonance Research (OCMR), Oxford, Oxfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No